CLINICAL TRIAL: NCT01607905
Title: A Phase I Study of the Safety, Pharmacokinetics and Pharmacodynamics of Escalating Doses of the Selective Inhibitor of Nuclear Export/SINE Compound KPT-330 in Patients With Advanced or Metastatic Solid Tumor Malignancies
Brief Title: Safety Study of KPT-330 (Selinexor) in Patients With Advanced or Metastatic Solid Tumor Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-002
Record Dates: First submitted 2012-05-16; First posted 2012-05-30 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor
Keywords: Selinexor; KPT-330; Squamous Cell Carcinoma; Glioblastoma multiforme; Adenocarcinoma; Melanoma; Colorectal cancer; Gynecological cancer; Castrate-resistant Prostate Cancer; Other solid tumors
MeSH Terms: conditions — Carcinoma, Squamous Cell; Glioblastoma; Adenocarcinoma; Melanoma; Colorectal Neoplasms | interventions — selinexor; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A (Colorectal Cancer) (Experimental): Participants with colorectal cancer and liver metastasis received oral selinexor as single agent in 8 schedules, Schedule1: ≤12milligrams per meter square(mg/m^2) 3 times weekly(TIW) during Weeks 1 and 3, twice weekly(BIW) during Weeks 2 and 4 up to 10 doses/cycle(28 days/cycle); Schedule2: >12mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle(28 days/cycle); Schedule3: ≥30mg/m^2 BIW(Days 1 and 3) up to 8 doses/cycle(28 days/cycle); Schedule4: ≥20mg/m^2 BIW(Days 1 and 2) up to 8 doses/cycle(28 days/cycle); Schedule5: ≥35mg/m^2 BIW(Days 1 and 4) up to 8 doses(28 days/cycle); Schedule6: ≥20mg/m^2 BIW(Days 1 and 4) after 500 mg(Week 1) to 1000 mg(Week 2 onwards) acetaminophen(given 1 hour prior to each selinexor dose) up to 8 doses/cycle (28 days/cycle); Schedule7: ≥50mg/m^2 once weekly(QW) up to 4 doses/cycle(28 days per cycle); Schedule8: ≥45mg/m^2 BIW(Days 1 and 3) up to 4 doses/cycle(21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor; Drug: Acetaminophen
- Arm B (Gynecological Cancer) (Experimental): Participants with gynecological cancer received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor
- Arm C (Squamous Cell Cancer) (Experimental): Participants with squamous cell cancer received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor
- Arm D (Castrate-resistant Prostate Cancer) (Experimental): Participants with castrate-resistant prostate cancer (CRPC) received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor
- Arm E (Glioblastoma Multiforme) (Experimental): Participants with glioblastoma multiforme (GBM) received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor
- Arm F (Melanoma) (Experimental): Participants with Melanoma received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor
- Arm G (Other Solid Tumors) (Experimental): Participants with other solid tumors received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Participants in this study will receive selinexor orally at dose levels specified for their respective dose cohorts. Dosing will begin at 3 mg/m^2 twice a week and will escalate until the MTD or RP2D is determined. Cycles will be repeated in 4-week (28 days for schedule 1 to 7) and 3-week (21 days for schedule 8) intervals until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, dose adjustment will be permitted.
  Other Names: KPT-330; XPOVIO
Drug: Acetaminophen — Oral 500 mg (in Cycle 1, Week 1) to 1000 mg (in Cycle 1, Week 2 and onwards) of acetaminophen will be administered 1 hour prior to each selinexor dose up to 8 doses per cycle (28 days per cycle)
  Arms: Arm A (Colorectal Cancer)

SUMMARY:
Phase 1 study to evaluate the safety and tolerability of selinexor and determine the Recommended Phase 2 Dose (RP2D) of selinexor for advanced or metastatic solid tumor malignancies.

DETAILED DESCRIPTION:
This is a phase 1a and phase 1b, open-label, dose-escalation study to evaluate the safety and tolerability of selinexor and determine the RP2D in patients with solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Dose Escalation Phase: Patients with advanced or metastatic solid tumors for which no standard therapy is available. For Schedule 6 only: patients with colorectal cancer with liver metastasis.

   Dose Expansion Phase: Previously treated, metastatic or advanced recurrent malignancy with 1 of the following diagnoses, which has been confirmed histologically or cytologically:
   * Up to 12 patients with metastatic colorectal cancer with a history of progression or recurrence following prior fluoropyrimidine, irinotecan and platinum containing regimens as well as bevacizumab. In addition, patients with Kras wild type tumor must have received at least one EGFR blocker.
   * Up to 6 patients with histological or cytological documentation of advanced ovarian, fallopian tube, or primary peritoneal carcinoma with a history of progression or recurrence following at least one prior platinum and one taxane based chemotherapy
   * Up to 12 patients with incurable Squamous cell cancers as follows:

     1. A minimum of 4 Squamous Non-Small Cell Lung Cancer (Sq-NSCLC)
     2. A minimum of 4 Squamous Cell Carcinomas of the Head and Neck (Sq-HNC)
     3. Squamous Cell Carcinoma of the Cervix (SqCC) All patient with Squamous Cell Carcinomas should have a documented history of progression or recurrence following at least one prior platinum based chemotherapy or chemotherapy/radiation containing regimen
   * Up to 6 patients with castration-resistant prostate cancer (CRPC) that was pathologically confirmed as adenocarcinoma of the prostate and with evidence of metastatic disease on bone scan or other imaging. Patient must have progressive disease after at least one hormonal treatment and one cytotoxic therapy e.g. with docetaxel, mitoxantrone.
   * Up to 12 patients with unresectable metastatic melanoma whose disease progressed on at least 1 prior systemic anticancer regimen (chemotherapy, biological or immunotherapy, or targeted therapy). Enrollment to this cohort may have been stopped before reaching 12 patients once the dose-escalation portion of the study was completed.
   * Approximately 6 patients with advanced or metastatic solid tumors were to be enrolled on Schedule 8 at a starting dose of 35 mg/m^2 to assess general tolerability and activity of selinexor.
2. Dose Escalation Phase: Patients have exhausted, or be deemed to not benefit from, further conventional therapy and have evidence of progressive disease on study entry.

Both Dose Escalation and Expansion Phases: There is no upper limit on the number of prior treatments provided that all inclusion criteria are met and exclusion criteria are not met. Hormone ablation therapy is considered an anticancer regimen. Radiation and surgery are not considered anticancer regimes.

Exclusion Criteria:

1. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤3 weeks prior to cycle 1 day 1 and mitomycin C and radioimmunotherapy 6 weeks prior to cycle 1 day 1;
2. Except for patients with GBM/ AnaA in the Expansion Phase, patients with active CNS malignancy are excluded. Asymptomatic small lesions are not considered active. Treated lesions may be considered inactive if they are stable for at least 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-06-18 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
- Princess Margaret Hospital, Toronto, Ontario, Canada
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Machlus KR, Wu SK, Vijey P, Soussou TS, Liu ZJ, Shacham E, Unger TJ, Kashyap T, Klebanov B, Sola-Visner M, Crochiere M, Italiano JE Jr, Landesman Y. Selinexor-induced thrombocytopenia results from inhibition of thrombopoietin signaling in early megakaryopoiesis. Blood. 2017 Aug 31;130(9):1132-1143. doi: 10.1182/blood-2016-11-752840. Epub 2017 Jun 19. PMID 28630120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at six centers in United States, Canada, and Denmark from 18 June 2012 and 15 March 2016.
Pre-assignment Details: A total of 192 participants were enrolled, of which 191 participants started study (1 participant reported missing malignancy), 189 participants received at least 1 dose of study drug.
Groups:
- Arm A (Colorectal Cancer): Participants with colorectal cancer with liver metastasis received oral selinexor as a single agent in eight schedules- Schedule 1: ≤12 milligrams per meter square (mg/m^2) 3 times weekly (TIW) during Weeks 1 and 3, twice weekly (BIW) during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW(Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 6: ≥20 mg/m^2 BIW (Days 1 and 4) after 500 mg (Cycle 1, Week 1) to 1000 mg (Cycle 1, Week 2 onwards) acetaminophen (given 1 hour prior to each selinexor dose) up to 8 doses/cycle(28 days/cycle); Schedule 7: ≥50 mg/m^2 once weekly (QW) up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
- Arm D (Castrate-resistant Prostate Cancer): Participants with CRPC received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
- Arm E (Glioblastoma Multiforme): Participants with GBM received oral selinexor as a single agent in eight schedules, Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW (Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Started | 60 | 20 | 21 | 21 | 7 | 15 | 47
Received Study Drug | 59 | 20 | 21 | 21 | 6 | 15 | 47
Low Dose (<30 mg/m^2) | 16 | 5 | 3 | 0 | 0 | 2 | 8
Medium Dose (>=30 mg/m^2 and <55 mg/m^2) | 27 | 11 | 15 | 8 | 6 | 3 | 21
High Dose (>= 55 mg/m^2) | 16 | 4 | 3 | 13 | 0 | 10 | 18
Completed (Participants who completed study treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 60 | 20 | 21 | 21 | 7 | 15 | 47
Not completed — Withdrawal by participant | 7 | 2 | 4 | 6 | 0 | 4 | 12
Not completed — Incidence or severity of AEs | 5 | 1 | 1 | 3 | 0 | 2 | 8
Not completed — Disease progression | 44 | 16 | 15 | 11 | 6 | 7 | 21
Not completed — Non-compliance with study procedures | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 1 | 1 | 1 | 1 | 0 | 0 | 3
Not completed — Other treatments become available | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Randomized but not treated | 1 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of selinexor. As pre-specified in the study Protocol data were not collected per dose level. The limited data available based on cancer stratification as pre-specified in the protocol is presented.
Groups:
- Arm A (Colorectal Cancer): Participants with colorectal cancer with liver metastasis received oral selinexor as a single agent in eight schedules- Schedule 1: ≤12 milligrams per meter square (mg/m^2) 3 times weekly (TIW) during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW(Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 6: ≥20 mg/m^2 BIW (Days 1 and 4) after 500 mg (Cycle 1, Week 1) to 1000 mg (Cycle 1, Week 2 onwards) acetaminophen (given 1 hour prior to each selinexor dose) up to 8 doses/cycle(28 days/cycle); Schedule 7: ≥50 mg/m^2 once weekly (QW) up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors) | Total
Number analyzed (Participants) | 59 | 20 | 21 | 21 | 6 | 15 | 47 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (11.35) | 55.0 (12.54) | 59.2 (7.39) | 68.7 (7.69) | 56.0 (14.94) | 67.7 (11.04) | 57.7 (12.67) | 60.2 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 9 | 0 | 3 | 4 | 14 | 75
  Male | 34 | 0 | 12 | 21 | 3 | 11 | 33 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 0 | 4 | 2 | 0 | 1 | 5 | 22
  White | 45 | 18 | 17 | 16 | 6 | 14 | 41 | 157
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAE was defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) was defined as an AE that meets one or more of the mentioned criteria; is fatal, life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly/birth defect, or important medical events. Number of participants with TEAEs and TESAEs were reported.
Time Frame: From start of study drug administration to 30 days after last dose of study treatment (maximum duration of 45 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Colorectal Cancer): Participants with colorectal cancer with liver metastasis received oral selinexor as a single agent in eight schedules- Schedule 1: ≤12 mg/m^2 TIW during Weeks 1 and 3, BIW during Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 2: >12 mg/m^2 TIW during Weeks 1 and 3, BIW in Weeks 2 and 4 up to 10 doses/cycle (28 days/cycle); Schedule 3: ≥30 mg/m^2 BIW(Days 1 and 3) up to 8 doses/cycle (28 days/cycle); Schedule 4: ≥20 mg/m^2 BIW (Days 1 and 2) up to 8 doses/cycle (28 days/cycle); Schedule 5: ≥35 mg/m^2 BIW (Days 1 and 4) up to 8 doses (28 days/cycle); Schedule 6: ≥20 mg/m^2 BIW (Days 1 and 4) after 500 mg (Cycle 1, Week 1) to 1000 mg (Cycle 1, Week 2 onwards) acetaminophen (given 1 hour prior to each selinexor dose) up to 8 doses/cycle(28 days/cycle); Schedule 7: ≥50 mg/m^2 QW up to 4 doses/cycle (28 days per cycle); Schedule 8: ≥45 mg/m^2 BIW (Days 1 and 3) up to 4 doses/cycle (21 days/cycle), until disease progression, death, or unacceptable toxicity.
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 59 | 20 | 21 | 21 | 6 | 15 | 47
Participants
  Participants with TEAEs | 59 | 20 | 21 | 21 | 6 | 15 | 46
  Participants with TESAEs | 30 | 13 | 9 | 8 | 2 | 5 | 24

2. Primary Outcome: Number of Participants With Treatment-related Treatment-emergent Adverse Events
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAE was defined as an adverse event with an onset that occurs after receiving study drug. A treatment-related AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product; the event had a causal relationship with the treatment or usage.
Time Frame: From start of study drug administration to 30 days after last dose of study treatment (maximum duration of 45 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 59 | 20 | 21 | 21 | 6 | 15 | 47
Participants
  Participants with Treatment-related TEAEs | 59 | 19 | 20 | 21 | 6 | 14 | 45
  Participants with Treatment-related TESAEs | 6 | 2 | 1 | 4 | 1 | 1 | 9

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Greater Than or Equal to Grade 3, Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE), Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. A treatment related AE was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event had a causal relationship with the treatment or usage.
Time Frame: From start of study drug administration to 30 days after last dose of study treatment (maximum duration of 45 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 59 | 20 | 21 | 21 | 6 | 15 | 47
Participants | 50 | 17 | 16 | 17 | 4 | 11 | 35

4. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicity (DLT)
Description: Evaluation of DLTs was only conducted in participants who participated in the Dose-escalation Phase. A DLT was defined as any of the following, considered possibly related to drug administration, occurring in the first 28 days (or 21 days for participants on Schedule 8) at the target dose (ie, for Schedule 2 this meant the first 4 weeks after the 12 mg/m2 run-in week): Missed selinexor doses due to drug-related toxicities, discontinuation of a participant due to a toxicity that was at least possibly related to study drug before completing Cycle 1.
Time Frame: Cycle 1 only (28-day cycle)
Population: DLT Evaluable Population included all participants enrolled to the study during the dose-escalation phase who met the inclusion/exclusion criteria on first day of dosing and completed at least 1 cycle of therapy or experienced a DLT during the first cycle. As pre-specified in the study Protocol data were not collected per dose level. The limited data available based on cancer stratification as pre-specified in the protocol is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 59 | 20 | 21 | 21 | 6 | 15 | 47
Participants | 1 | 0 | 0 | 0 | 0 | 1 | 2

5. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The RP2D was the maximum tolerated dose (MTD) or less. MTD was defined as the next lower dose level below the one in which >1 of 3 participants or ≥2 of 6 participants experienced DLT, provided that dose level was ≤25 percent (%) lower than the highest (intolerable) dose tested. If the projected MTD was >25% lower than the highest dose tested, then an additional cohort of ≥3 participants was added at a dose that was intermediate between the intolerable dose and the next lower dose.
Time Frame: From start of study drug administration to 30 days after last dose of study treatment (maximum duration of 45 months)
Population: Safety Population included all participants who received at least one dose of selinexor. The data in terms of dose was reported as combined data for participants from all arms, pre-specified in protocol. Here, 'Overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Number; unit: mg/m^2
Groups:
- Arms A to G: Overall Solid Tumor Malignancies: Participants with colorectal cancer with liver metastasis, gynecological cancer, squamous cell cancer, CRPC, GBM, melanoma, other solid tumors received oral selinexor as a single agent in eight schedules, schedule 1. ≤12 mg/m^2 TIW in Weeks 1 and 3, BIW in Weeks 2 and 4, schedule 2. >12 mg/m^2 TIW in Weeks 1 and 3, BIW in Weeks 2 and 4, schedule 3. ≥ 30 mg/m^2 BIW (Days 1 and 3), schedule 4. ≥20 mg/m^2 BIW (Days 1 and 2), schedule 5. ≥35 mg/m^2 BIW (Days 1 and 4), schedule 6. ≥20 mg/m^2 BIW (Days 1 and 4), schedule 7. ≥50 mg/m^2 once weekly (QW), schedule 8. ≥45 mg/m^2 BIW (Days 1 and 3) until disease progression, death, or unacceptable toxicity.
Arm/Group | Arms A to G: Overall Solid Tumor Malignancies
Number analyzed (Participants) | 82
mg/m^2 | 35

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Selinexor
Description: Cmax was defined as maximum observed concentration, taken directly from the plasma concentration data.
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: Pharmacokinetic (PK) population consisted of all participants who received selinexor, and had evaluable PK for at least one dosing occasion. Data for the PK parameters were planned and analyzed based on doses and % coefficient of variation was not evaluable for arms where single participant was analyzed. Here, 'Overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Groups:
- Selinexor Dose: 3 mg/m^2: Participants received 3 milligram per square meter (mg/m^2) of selinexor for Cycle1 Day1.
- Selinexor Dose: 6 mg/m^2: Participants received single oral dose of 6 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 12 mg/m^2: Participants received single oral dose of 12 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 16.8 mg/m^2: Participants received single oral dose of 16.8 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 20 mg/m^2: Participants received single oral dose of 20 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 23 mg/m^2: Participants received single oral dose of 23 mg/m^2 Selinexor for Cycle1Day1.
- Selinexor Dose: 28 mg/m^2: Participants received single oral dose of 28 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 30 mg/m^2: Participants received single oral dose of 30 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 35 mg/m^2: Participants received single oral dose of 35 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 39 mg/m^2: Participants received single oral dose of 39 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 40 mg/m^2: Participants received single oral dose of 40 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 45 mg/m^2: Participants received single oral dose of 45 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 50 mg/m^2: Participants received single oral dose of 50 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 55 mg/m^2: Participants received single oral dose of 55 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 58 mg/m^2: Participants received single oral dose of 58 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 65 mg/m^2: Participants received single oral dose of 65 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 70 mg/m^2: Participants received single oral dose of 70 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 80 mg/m^2: Participants received single oral dose of 80 mg/m^2 Selinexor for Cycle1 Day1.
- Selinexor Dose: 85 mg/m^2: Participants received single oral dose of 85 mg/m^2 Selinexor for Cycle1 Day1.
Arm/Group | Selinexor Dose: 3 mg/m^2 | Selinexor Dose: 6 mg/m^2 | Selinexor Dose: 12 mg/m^2 | Selinexor Dose: 16.8 mg/m^2 | Selinexor Dose: 20 mg/m^2 | Selinexor Dose: 23 mg/m^2 | Selinexor Dose: 28 mg/m^2 | Selinexor Dose: 30 mg/m^2 | Selinexor Dose: 35 mg/m^2 | Selinexor Dose: 39 mg/m^2 | Selinexor Dose: 40 mg/m^2 | Selinexor Dose: 45 mg/m^2 | Selinexor Dose: 50 mg/m^2 | Selinexor Dose: 55 mg/m^2 | Selinexor Dose: 58 mg/m^2 | Selinexor Dose: 65 mg/m^2 | Selinexor Dose: 70 mg/m^2 | Selinexor Dose: 80 mg/m^2 | Selinexor Dose: 85 mg/m^2
Number analyzed (Participants) | 1 | 3 | 7 | 1 | 5 | 5 | 8 | 16 | 10 | 4 | 6 | 3 | 4 | 3 | 4 | 7 | 1 | 2 | 3
nanogram per milliliter | 30 | 75 (38.2) | 149 (32) | 168 | 220 (44.5) | 308 (12.1) | 293 (58.3) | 413 (46.7) | 349 (25.4) | 528 (12.5) | 442 (63.6) | 390 (25.3) | 507 (57.8) | 505 (18.2) | 561 (45.4) | 896 (71.7) | 521 | 765 (6.6) | 1371 (31.1)

7. Secondary Outcome: Time of Maximum Observed Concentration in Plasma (Tmax) of Selinexor
Description: Tmax was defined as time of first observation of Cmax, taken directly from the plasma concentration data.
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: PK population consisted of all participants who received selinexor, and had evaluable PK for at least one dosing occasion. Data for the PK parameters were planned and analyzed based on doses and full range data was not evaluable for arms with single participant. Here, 'Overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Median (Full Range); unit: hours
Groups:
- Selinexor Dose: 3 mg/m^2: Participants received 3 mg/m^2 of selinexor for Cycle1 Day1.
- Selinexor Dose: 23 mg/m^2: Participants received single oral dose of 23 mg/m^2 Selinexor for Cycle1 Day1.
Arm/Group | Selinexor Dose: 3 mg/m^2 | Selinexor Dose: 6 mg/m^2 | Selinexor Dose: 12 mg/m^2 | Selinexor Dose: 16.8 mg/m^2 | Selinexor Dose: 20 mg/m^2 | Selinexor Dose: 23 mg/m^2 | Selinexor Dose: 28 mg/m^2 | Selinexor Dose: 30 mg/m^2 | Selinexor Dose: 35 mg/m^2 | Selinexor Dose: 39 mg/m^2 | Selinexor Dose: 40 mg/m^2 | Selinexor Dose: 45 mg/m^2 | Selinexor Dose: 50 mg/m^2 | Selinexor Dose: 55 mg/m^2 | Selinexor Dose: 58 mg/m^2 | Selinexor Dose: 65 mg/m^2 | Selinexor Dose: 70 mg/m^2 | Selinexor Dose: 80 mg/m^2 | Selinexor Dose: 85 mg/m^2
Number analyzed (Participants) | 1 | 3 | 7 | 1 | 5 | 5 | 8 | 16 | 10 | 4 | 6 | 3 | 4 | 3 | 4 | 7 | 1 | 2 | 3
hours | 1 | 2.1 [0.9 to 7.5] | 2.0 [1.0 to 7.7] | 2.1 | 2.3 [2.0 to 7.5] | 2.1 [1.1 to 8.0] | 3.1 [0.5 to 7.6] | 2.9 [0.5 to 7.7] | 3.8 [2.0 to 7.8] | 3.1 [1.0 to 4.3] | 3.9 [2.1 to 4.2] | 4.2 [2.1 to 8.0] | 3.0 [1.0 to 4.1] | 3.8 [1.1 to 4.0] | 3.1 [2.2 to 4.2] | 2.0 [0.6 to 7.5] | 8.0 | 3.9 [3.8 to 4.0] | 3.9 [3.8 to 3.9]

8. Secondary Outcome: Area Under the Concentration Time Curve From the Time of Dosing to Time in Plasma (AUC0-t) of Selinexor
Description: AUC0-t was defined as area under the concentration-time curve from time zero to the last non-zero concentration.
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: PK population consisted of all participants who received selinexor, and had evaluable PK for at least one dosing occasion. Data for the PK parameters were planned and analyzed based on doses and % coefficient of variation was not evaluable for arms with single participant. Here, 'Overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter
Arm/Group | Selinexor Dose: 3 mg/m^2 | Selinexor Dose: 6 mg/m^2 | Selinexor Dose: 12 mg/m^2 | Selinexor Dose: 16.8 mg/m^2 | Selinexor Dose: 20 mg/m^2 | Selinexor Dose: 23 mg/m^2 | Selinexor Dose: 28 mg/m^2 | Selinexor Dose: 30 mg/m^2 | Selinexor Dose: 35 mg/m^2 | Selinexor Dose: 39 mg/m^2 | Selinexor Dose: 40 mg/m^2 | Selinexor Dose: 45 mg/m^2 | Selinexor Dose: 50 mg/m^2 | Selinexor Dose: 55 mg/m^2 | Selinexor Dose: 58 mg/m^2 | Selinexor Dose: 65 mg/m^2 | Selinexor Dose: 70 mg/m^2 | Selinexor Dose: 80 mg/m^2 | Selinexor Dose: 85 mg/m^2
Number analyzed (Participants) | 1 | 3 | 7 | 1 | 5 | 5 | 8 | 16 | 10 | 4 | 6 | 3 | 4 | 3 | 4 | 7 | 1 | 2 | 3
nanogram hour per milliliter | 333 | 707 (13.6) | 1578 (21.0) | 1369 | 2446 (23.3) | 3387 (17.7) | 3106 (31) | 3861 (16.6) | 3691 (25.0) | 4885 (15.3) | 5255 (24.4) | 4390 (24.9) | 5490 (3.1) | 5803 (23.5) | 5888 (18.9) | 8482 (44.8) | 7210 | 9838 (12.7) | 11485 (20.1)

9. Secondary Outcome: Area Under the Concentration Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of Selinexor
Description: AUC0-inf was defined as area under the concentration-time curve from time zero to infinity (extrapolated). It was calculated as AUC0-t + Ct/kel, where: Ct = the last observed non-zero concentration and Kel = elimination rate constant.
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter
Arm/Group | Selinexor Dose: 3 mg/m^2 | Selinexor Dose: 6 mg/m^2 | Selinexor Dose: 12 mg/m^2 | Selinexor Dose: 16.8 mg/m^2 | Selinexor Dose: 20 mg/m^2 | Selinexor Dose: 23 mg/m^2 | Selinexor Dose: 28 mg/m^2 | Selinexor Dose: 30 mg/m^2 | Selinexor Dose: 35 mg/m^2 | Selinexor Dose: 39 mg/m^2 | Selinexor Dose: 40 mg/m^2 | Selinexor Dose: 45 mg/m^2 | Selinexor Dose: 50 mg/m^2 | Selinexor Dose: 55 mg/m^2 | Selinexor Dose: 58 mg/m^2 | Selinexor Dose: 65 mg/m^2 | Selinexor Dose: 70 mg/m^2 | Selinexor Dose: 80 mg/m^2 | Selinexor Dose: 85 mg/m^2
Number analyzed (Participants) | 1 | 2 | 5 | 1 | 3 | 4 | 1 | 10 | 4 | 3 | 6 | 1 | 2 | 3 | 2 | 5 | 0 | 1 | 2
nanogram hour per milliliter | 355 | 808 (5.2) | 1613 (21.4) | 1455 | 2269 (27.2) | 3332 (17.3) | 3936 | 3961 (12.1) | 4585 (18.2) | 5014 (18.0) | 5294 (24.0) | 3395 | 5688 (0.6) | 5894 (24.8) | 6567 (12.8) | 10265 (31.4) |  | 9025 | 11830 (20.1)

10. Secondary Outcome: Elimination Half-Life (t1/2) of Selinexor
Description: t1/2 was defined as elimination half-life, it was calculated as ln(2)/kel, where In = natural logarithm and kel = elimination rate constant.
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: PK population consisted of all participants who received selinexor, and had evaluable PK for at least one dosing occasion. Data for the PK parameters were planned and analyzed based on doses and full range was not evaluable for arms with single participant. Here, 'Overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Selinexor Dose: 3 mg/m^2 | Selinexor Dose: 6 mg/m^2 | Selinexor Dose: 12 mg/m^2 | Selinexor Dose: 16.8 mg/m^2 | Selinexor Dose: 20 mg/m^2 | Selinexor Dose: 23 mg/m^2 | Selinexor Dose: 28 mg/m^2 | Selinexor Dose: 30 mg/m^2 | Selinexor Dose: 35 mg/m^2 | Selinexor Dose: 39 mg/m^2 | Selinexor Dose: 40 mg/m^2 | Selinexor Dose: 45 mg/m^2 | Selinexor Dose: 50 mg/m^2 | Selinexor Dose: 55 mg/m^2 | Selinexor Dose: 58 mg/m^2 | Selinexor Dose: 65 mg/m^2 | Selinexor Dose: 70 mg/m^2 | Selinexor Dose: 80 mg/m^2 | Selinexor Dose: 85 mg/m^2
Number analyzed (Participants) | 1 | 2 | 5 | 1 | 3 | 4 | 1 | 10 | 4 | 3 | 6 | 1 | 2 | 3 | 3 | 5 | 0 | 1 | 2
hours | 6.2 | 5.6 [4.8 to 6.4] | 5.0 [4.1 to 7.8] | 5.7 | 5.6 [4.2 to 7.5] | 5.8 [5.7 to 6.4] | 5.7 | 6.5 [4.1 to 7.9] | 6.0 [4.0 to 7.0] | 5.9 [3.5 to 6.2] | 6.9 [5.4 to 7.2] | 7.3 | 7.3 [7.1 to 7.5] | 6.2 [5.0 to 10.1] | 6.5 [5.6 to 7.1] | 6.9 [5.5 to 9.3] |  | 5.7 | 5.3 [4.6 to 6.0]

11. Secondary Outcome: Apparent Total Body Clearance (CL/F) of Selinexor
Description: CL/F was calculated as Dose/AUC0-inf, uncorrected for fraction absorbed; reported normalized by participant body weight (kilogram).
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour per kilogram
Groups:
- Selinexor Dose: 30 mg/m^2: Participants received single oral dose of 30 mg/m^2 Selinexor for Cycle1Day1.
Arm/Group | Selinexor Dose: 3 mg/m^2 | Selinexor Dose: 6 mg/m^2 | Selinexor Dose: 12 mg/m^2 | Selinexor Dose: 16.8 mg/m^2 | Selinexor Dose: 20 mg/m^2 | Selinexor Dose: 23 mg/m^2 | Selinexor Dose: 28 mg/m^2 | Selinexor Dose: 30 mg/m^2 | Selinexor Dose: 35 mg/m^2 | Selinexor Dose: 39 mg/m^2 | Selinexor Dose: 40 mg/m^2 | Selinexor Dose: 45 mg/m^2 | Selinexor Dose: 50 mg/m^2 | Selinexor Dose: 55 mg/m^2 | Selinexor Dose: 58 mg/m^2 | Selinexor Dose: 65 mg/m^2 | Selinexor Dose: 70 mg/m^2 | Selinexor Dose: 80 mg/m^2 | Selinexor Dose: 85 mg/m^2
Number analyzed (Participants) | 1 | 2 | 5 | 1 | 3 | 4 | 1 | 10 | 4 | 3 | 6 | 1 | 2 | 3 | 3 | 5 | 0 | 1 | 2
liter per hour per kilogram | 0.20 | 0.18 (7.9) | 0.19 (16) | 0.20 | 0.19 (27) | 0.19 (26.1) | 0.18 | 0.17 (16.8) | 0.20 (26.7) | 0.20 (12.5) | 0.19 (24.4) | 0.27 | 0.18 (10.6) | 0.20 (17.1) | 0.20 (17.0) | 0.15 (32.7) |  | 0.22 | 0.18 (4.1)

12. Secondary Outcome: Apparent Volume of Distribution of Selinexor (Vd/F)
Description: Vd/F was calculated as Dose/(kel * AUC0-inf), uncorrected for fraction absorbed; reported normalized by participant body weight (kilogram).
Time Frame: Cycle1, Day1: Pre-dose, 30, 60, 120, 240, 480 minutes
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per kilogram
Groups:
- Selinexor Dose: 3 Milligram Per Square Meter (mg/m2): Participants received 3 mg/m2 of selinexor for Cycle1Day1.
- Selinexor Dose: 6 mg/m2: Participants received single oral dose of 6 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 12 mg/m2: Participants received single oral dose of 12 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 16.8 mg/m2: Participants received single oral dose of 16.8 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 20 mg/m2: Participants received single oral dose of 20 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 23 mg/m2: Participants received single oral dose of 23 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 28 mg/m2: Participants received single oral dose of 28 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 30 mg/m2: Participants received single oral dose of 30 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 35 mg/m2: Participants received single oral dose of 35 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 39 mg/m2: Participants received single oral dose of 39 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 40 mg/m2: Participants received single oral dose of 40 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 45 mg/m2: Participants received single oral dose of 45 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 50 mg/m2: Participants received single oral dose of 50 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 55 mg/m2: Participants received single oral dose of 55 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 58 mg/m2: Participants received single oral dose of 58 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 65 mg/m2: Participants received single oral dose of 65 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 70 mg/m2: Participants received single oral dose of 70 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 80 mg/m2: Participants received single oral dose of 80 mg/m2 Selinexor for Cycle1Day1.
- Selinexor Dose: 85 mg/m2: Participants received single oral dose of 85 mg/m2 Selinexor for Cycle1Day1.
Arm/Group | Selinexor Dose: 3 Milligram Per Square Meter (mg/m2) | Selinexor Dose: 6 mg/m2 | Selinexor Dose: 12 mg/m2 | Selinexor Dose: 16.8 mg/m2 | Selinexor Dose: 20 mg/m2 | Selinexor Dose: 23 mg/m2 | Selinexor Dose: 28 mg/m2 | Selinexor Dose: 30 mg/m2 | Selinexor Dose: 35 mg/m2 | Selinexor Dose: 39 mg/m2 | Selinexor Dose: 40 mg/m2 | Selinexor Dose: 45 mg/m2 | Selinexor Dose: 50 mg/m2 | Selinexor Dose: 55 mg/m2 | Selinexor Dose: 58 mg/m2 | Selinexor Dose: 65 mg/m2 | Selinexor Dose: 70 mg/m2 | Selinexor Dose: 80 mg/m2 | Selinexor Dose: 85 mg/m2
Number analyzed (Participants) | 1 | 2 | 5 | 1 | 3 | 4 | 1 | 10 | 4 | 3 | 6 | 1 | 2 | 3 | 3 | 5 | 0 | 1 | 2
liter per kilogram | 1.8 | 1.4 (12.5) | 1.4 (22.5) | 1.6 | 1.6 (20.9) | 1.6 (21.2) | 1.5 | 1.6 (6.6) | 1.6 (26.6) | 1.5 (26.1) | 1.9 (31.1) | 2.8 | 1.9 (14.3) | 1.9 (24.7) | 1.8 (15.4) | 1.5 (31.8) |  | 1.8 | 1.4 (22.7)

13. Secondary Outcome: Number of Participants With Best Overall Response (BOR)
Description: BOR is response recorded from start of treatment until disease progression/recurrence. Best lesion response was defined by Recist Criteria V1 (for target and non-target lesions) and RANO criteria (for glioblastoma multiforme): complete response (CR)- disappearance of all target lesions. Any pathological lymph nodes (target/non target) must have reduction in short axis to less than (<) 10 mm; partial response (PR)- at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum longest diameter; stable disease (SD)- steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; progressive disease (PD): at least 20% increase in sum of diameters of measured lesions taking as references smallest sum of diameters recorded since treatment started. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm, or appearance of one or more new lesions.
Time Frame: Up to maximum duration of 45 months
Population: Efficacy Population included all participants registered to the study who had either completed 1 cycle of treatment or discontinued treatment prior to completing the first cycle due to documented disease progression, death related to disease, or treatment-related toxicity. As pre-specified in the study Protocol data were not collected per dose level. The limited data available based on cancer stratification as pre-specified in the protocol is presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 57 | 20 | 21 | 19 | 6 | 14 | 46
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Partial Response | 1 | 3 | 0 | 0 | 0 | 1 | 1
  Stable Disease | 15 | 9 | 5 | 11 | 0 | 3 | 20
  Progression (Objective) | 28 | 6 | 8 | 5 | 5 | 4 | 10
  Progressive Disease due to symptomatic deterioration | 4 | 0 | 3 | 0 | 0 | 1 | 1
  Not Evaluable | 9 | 2 | 5 | 3 | 1 | 4 | 14

14. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective response rate (ORR) was determined as percentage of participants who had either CR or PR, as defined by RECIST v1.1 (for solid tumors). CR was defined as disappearance of all target lesions. Any pathological lymph nodes (target/non target) must have reduction in short axis to <10 mm and PR was defined as at least 30% decrease in sum of diameters of target lesions. ORR was calculated as a proportion and included a 2 sided 95% CI using the exact (Clopper-Pearson) method.
Time Frame: Up to maximum duration of 45 months
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 57 | 20 | 21 | 19 | 6 | 14 | 46
percentage of participants | 1.8 | 15.0 | 0 | 0 | 0 | 14.3 | 2.2

15. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of stable disease was defined as the time from the date of first dose to first documented radiologic evidence of disease recurrence or progression, as defined by RECIST v1.1 (for solid tumors) or RANO criteria (for GBM and AnaA).
Time Frame: From first dose of study drug administration to first documented evidence of disease recurrence or progression (maximum duration of 45 months)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 57 | 20 | 21 | 19 | 6 | 14 | 46
Days | 53 [52 to 59] | 119 [42 to 310] | 52 [46 to 79] | 133 [53 to 484] | 43 [38 to 55] | 52 [22 to 539] | 134 [53 to 267]

16. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was calculated from the date of first dose of study treatment to first documented evidence of disease recurrence or progression or death due to any cause. Patients who are last known to be alive and without evidence of progression will be censored at time of last evaluable disease assessment. If date of progression or death occurred after more than 1 missed disease assessment interval, patients are censored at the time of last evaluable disease assessment prior to the missed assessment. Progressive disease was defined as at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded since the treatment started. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions also constituted progressive disease.
Time Frame: From start of study drug administration until PD or discontinuation from the study or death (maximum duration of 45 months)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 57 | 20 | 21 | 19 | 6 | 14 | 46
Days | 53 [52 to 59] | 119 [42 to 310] | 52 [44 to 79] | 127 [53 to 322] | 41 [38 to 55] | 52 [22 to 539] | 88 [53 to 234]

17. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from the date of first dose to date of death. Participants who were still alive prior to the data cutoff for final efficacy analysis, or who dropout prior to study end, were censored at the day they were last known to be alive. The OS was calculated using the Kaplan-Meier method.
Time Frame: From first dose of study drug administration to date of death (maximum duration of 45 months)
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Number analyzed (Participants) | 57 | 20 | 21 | 19 | 6 | 14 | 46
Days | 136 [102 to 532] | 491 [167 to NA] — Here, 'NA' signifies that data was not evaluable for specific arms as the model can't estimate the data when the death events during the study was less than 50%. | 161 [62 to 460] | 354 [322 to NA] — Here, 'NA' signifies that data was not evaluable for specific arms as the model can't estimate the data when the death events during the study was less than 50%. | 103 [38 to 152] | NA [125 to NA] — Here, 'NA' signifies that data was not evaluable for specific arms as the model can't estimate the data when the death events during the study was less than 50%. | 290 [263 to NA] — Here, 'NA' signifies that data was not evaluable for specific arms as the model can't estimate the data when the death events during the study was less than 50%.

ADVERSE EVENTS:
Time Frame: From start of study drug administration to 30 days after last dose of study treatment (maximum duration of 45 months)
Description: As pre-specified in the study Protocol data were not collected per dose level. The limited data available based on cancer stratification as pre-specified in the protocol is presented.
Arm/Group | Arm A (Colorectal Cancer) | Arm B (Gynecological Cancer) | Arm C (Squamous Cell Cancer) | Arm D (Castrate-resistant Prostate Cancer) | Arm E (Glioblastoma Multiforme) | Arm F (Melanoma) | Arm G (Other Solid Tumors)
Serious Adverse Events (participants affected / at risk) | 30/59 | 13/20 | 9/21 | 8/21 | 2/6 | 5/15 | 24/47
Other Adverse Events (participants affected / at risk) | 59/59 | 20/20 | 21/21 | 21/21 | 6/6 | 15/15 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Colorectal Cancer) (N=59) | Arm B (Gynecological Cancer) (N=20) | Arm C (Squamous Cell Cancer) (N=21) | Arm D (Castrate-resistant Prostate Cancer) (N=21) | Arm E (Glioblastoma Multiforme) (N=6) | Arm F (Melanoma) (N=15) | Arm G (Other Solid Tumors) (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Colorectal Cancer) (N=59) | Arm B (Gynecological Cancer) (N=20) | Arm C (Squamous Cell Cancer) (N=21) | Arm D (Castrate-resistant Prostate Cancer) (N=21) | Arm E (Glioblastoma Multiforme) (N=6) | Arm F (Melanoma) (N=15) | Arm G (Other Solid Tumors) (N=47)
Anaemia (Blood and lymphatic system disorders) | 23 (23) | 13 (13) | 13 (13) | 10 (10) | 3 (3) | 4 (4) | 21 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 (26) | 6 (6) | 9 (9) | 12 (12) | 3 (3) | 8 (8) | 23 (23)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 3 (3) | 8 (8) | 1 (1) | 4 (4) | 9 (9)
Leukopenia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 3 (3) | 4 (4) | 1 (1) | 4 (4) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 9 (9) | 7 (7) | 4 (4) | 8 (8) | 2 (2) | 3 (3) | 8 (8)
Cataract (Eye disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Periorbital oedema (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Photopsia (Eye disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 46 (46) | 19 (19) | 12 (12) | 9 (9) | 3 (3) | 11 (11) | 38 (38)
Vomiting (Gastrointestinal disorders) | 35 (35) | 17 (17) | 11 (11) | 7 (7) | 2 (2) | 5 (5) | 27 (27)
Constipation (Gastrointestinal disorders) | 21 (21) | 9 (9) | 6 (6) | 11 (11) | 1 (1) | 5 (5) | 22 (22)
Diarrhoea (Gastrointestinal disorders) | 24 (24) | 11 (11) | 8 (8) | 7 (7) | 1 (1) | 7 (7) | 16 (16)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 9 (9) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 17 (17)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 6 (6) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral mucosa haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 46 (46) | 16 (16) | 14 (14) | 17 (17) | 5 (5) | 10 (10) | 36 (36)
Pyrexia (General disorders) | 14 | 5 | 5 | 1 | 2 | 1 | 9
Oedema peripheral (General disorders) | 12 (12) | 5 (5) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 6 (6)
Chills (General disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Face oedema (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Lung infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural anxiety (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 32 (32) | 8 (8) | 11 (11) | 10 (10) | 4 (4) | 7 (7) | 19 (19)
Blood creatinine increased (Investigations) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 9 (9)
Blood alkaline phosphatase increased (Investigations) | 12 (12) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 9 (9) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
White blood cell count decreased (Investigations) | 4 (4) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 8 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lipase increased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Amylase increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood urea increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 42 (42) | 13 (13) | 11 (11) | 14 (14) | 5 (5) | 9 (9) | 33 (33)
Hyponatraemia (Metabolism and nutrition disorders) | 36 (36) | 8 (8) | 7 (7) | 6 (6) | 1 (1) | 9 (9) | 17 (17)
Dehydration (Metabolism and nutrition disorders) | 17 (17) | 6 (6) | 4 (4) | 8 (8) | 2 (2) | 1 (1) | 11 (11)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (16) | 6 (6) | 4 (4) | 5 (5) | 2 (2) | 1 (1) | 9 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (14) | 1 (1) | 2 (2) | 8 (8) | 3 (3) | 1 (1) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (13) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 9 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (8) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 9 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 20 (20) | 6 (6) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 14 (14)
Dizziness (Nervous system disorders) | 13 (13) | 7 (7) | 3 (3) | 7 (7) | 2 (2) | 3 (3) | 15 (15)
Headache (Nervous system disorders) | 10 (10) | 7 (7) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 12 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (9) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coital bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 9 (9) | 4 (4) | 9 (9) | 1 (1) | 3 (3) | 19 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (6) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 13 (13)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Koilonychia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immobile (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Embolism (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infarction (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes